CLINICAL TRIAL: NCT07048093
Title: Development of Standard Guidelines for Relaxation Exercises in Patients With Chronic Neck Pain and Determination of Their Effectiveness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Utku Berberoğlu, Assistant Proffesor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G.O. 2024/153
Record Dates: First submitted 2025-06-14; First posted 2025-07-02 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Non Specific Chronic Neck Pain
Keywords: Relaxation Exercise; craniocervical flexion; upper trapezius
MeSH Terms: interventions — Exercise; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation Exercises Group (Experimental): This group will do relaxation exercises based on reciprocal inhibition, autogenic inhibition, proprioceptive training and postural training.
  Interventions: Other: Exercise
- Just Lie Back Group (Sham Comparator): This group do nothing but just lie back before and after actual measurements.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Other: Exercise — Average of 10 minutes relaxation exercises guided with a standard audio record based on reciprocal and autogenic muscle inhibition, proprioceptive training and postural training.
  Arms: Relaxation Exercises Group
Other: Sham (No Treatment) — This group take no treatment between actual before and after measurements.
  Arms: Just Lie Back Group

SUMMARY:
The goal of this observational study is to determine whether relaxation exercises performed before cranio-cervical flexion can reduce superficial neck muscle activation (specifically sternocleidomastoid and upper trapezius) in individuals with neck pain.

The main questions it aims to answer are:

* Does performing relaxation exercises prior to cranio-cervical flexion reduce sternocleidomastoid (SCM) muscle activation?
* Does it reduce upper trapezius muscle activation during the standing?

Researchers will compare the group performing relaxation exercises before cranio-cervical flexion to the group performing only cranio-cervical flexion to see if there is a measurable difference in superficial neck muscle activation.

Participants will:

* Perform cranio-cervical flexion exercises.
* Perform relaxation exercises prior to the cranio-cervical flexion (intervention group only).
* Undergo surface EMG measurements to assess muscle activity.

ELIGIBILITY:
Inclusion Criteria:

* Knowledge of Turkish
* Chronic (at least three months) neck pain
* Neck pain level of 4 or higher on a numerical pain scale

Exclusion Criteria:

* Neck pain caused by a tumor, trauma, or rheumatic disease
* History of surgery involving the head, neck, shoulder, or thoracic region
* Root compression
* Regular use of painkillers due to another illness
* Another illness severe enough to interfere with work

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | At enrollment (pre-intervention) and immediately after the relaxation exercise intervention or sham intervention (Day 1)
  On the numerical pain scale, the patient will be asked, "0 means no pain at all, 10 means unbearable pain, representing the worst pain/unbearable pain you have ever experienced. On a scale of 0 to 10, how would you rate your pain?"
Turkish Version of Core Outcome Measure Index for Neck Pain | At enrollment (pre-intervention)
  The first question consists of two 10-point numerical pain scales that ask about neck and arm-shoulder pain. Whichever of these two questions receives a higher response is used. The other five questions are five point Likert-type response questions. The six items cover five dimensions: pain intensity (neck and arm/shoulder pain), neck-related function, symptom-specific well-being, overall quality of life, and disability (social and work). The total score is calculated by taking the average of all responses. To form the Core Outcome Measure Index summary score, each of the dimension scores is transformed to a 0-10 scale and these are then averaged to give a score ranging from 0 to 10, with higher scores indicating a worse status.
EMG Activation Level of Sternocleidomastoid Muscle During Craniocervical Flexion Maneuver | At enrollment (pre-intervention) and immediately after the relaxation exercise intervention (Day 1)
  EMG Activation Level of Sternocleidomastoid Muscle During Craniocervical Flexion Maneuver standardized with Stabilizer Pressure Biofeedback Device
EMG Activation Level of Upper Trapezius Muscle During Standing Still | At enrollment (pre-intervention) and immediately after the relaxation exercise intervention (Day 1)
  EMG Activation Level of Upper Trapezius Muscle During Standing Still

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Balıkesir, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
This ethics committee has not yet established a data policy regarding open data. Otherwise, I would share it once it has been anonymised. I am still discussing this matter with the committee.

REFERENCES:
- [Background] Rota E, Evangelista A, Ceccarelli M, Ferrero L, Milani C, Ugolini A, Mongini F. Efficacy of a workplace relaxation exercise program on muscle tenderness in a working community with headache and neck pain: a longitudinal, controlled study. Eur J Phys Rehabil Med. 2016 Aug;52(4):457-65. Epub 2016 Jan 8. PMID 26745361
- [Background] Lee BK, Seo DK. The Importance of Optimal Gaze Direction on Deep Neck Flexor Activation in Chronic Neck Pain. Healthcare (Basel). 2020 Nov 1;8(4):449. doi: 10.3390/healthcare8040449. PMID 33139645
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880